CLINICAL TRIAL: NCT07000227
Title: Mechanism of FODMAP Restriction on Gut Microbiota and Gut Barrier Function in Functional Gastrointestinal Disorder Patients : A Randomised Controlled Trial
Brief Title: Mechanism of FODMAP Restriction on FGID Patients
Acronym: BRIDGE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Principal Investigator, Dr Shanthi Krishnasamy, Assistant Professor, Universiti Kebangsaan Malaysia Medical Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JEP-2024-1144; FRGS/1/2023/SKK06/UKM/03/4 (Other Grant/Funding Number: Ministry of Higher Education Malaysia)
Record Dates: First submitted 2025-05-05; First posted 2025-06-02 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Functional Gastrointestinal Disorders (FGIDs); Irritable Bowel Syndrome (IBS); Functional Dyspepsia
Keywords: Functional Gastrointestinal Disorder; Irritable Bowel Syndrome; Functional Dyspepsia; FODMAP Restriction; Gentle FODMAP
MeSH Terms: conditions — Gastrointestinal Diseases; Irritable Bowel Syndrome | interventions — FODMAP Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low FODMAP diet (Active Comparator): Low FODMAP diet will be administered for two weeks
  Interventions: Behavioral: Low FODMAP diet
- Gentle FODMAP diet (Active Comparator): Gentle FODMAP diet will be administered for two weeks
  Interventions: Behavioral: Gentle FODMAP diet
- Traditional Dietary Advice (Active Comparator): Traditional Dietary advice will be administered for two weeks
  Interventions: Behavioral: Traditional Dietary Advice

INTERVENTIONS:
Behavioral: Low FODMAP diet — High FODMAP foods are swapped for low FODMAP alternatives, for two weeks (Elimination phase)
  Arms: Low FODMAP diet
Behavioral: Gentle FODMAP diet — Key High FODMAP foods will be identified from patients' food diaries and swapped with low FODMAP alternatives. (Elimination phase)
  Arms: Gentle FODMAP diet
Behavioral: Traditional Dietary Advice — Subjects are required to follow a set of healthy eating guidelines set by NICE guidelines for IBS for two weeks a. Have regular meals and take time to eat b. Avoid missing meals or leaving long gaps between eating c. Drink at least eight cups of fluid a day, especially water or other non-d. caffeinated drinks, such as herbal teas d. Restrict tea and coffee to three cups a day e. Reduce intake of alcohol and fizzy drinks . Limit intake of high-fibre food g. Reduce intake of resistant starch h. Limit fresh fruit to three portions a day
  Arms: Traditional Dietary Advice

SUMMARY:
Brief Summary :

The goal of this clinical trial is to investigate the effects of differing FODMAP diets on gut microbiota, gut barrier function, symptom severity, quality of life, and psychological status in FGID patients. The main question it aims to answer is :

How does diets with differing FODMAP content affect the gut microbiota, gut barrier function, symptom severity, psychological status and quality of life in patients with FGID ? Researchers will compare low FODMAP diet, Gentle FODMAP diet and Traditional Dietary Advice (NICE guidelines) to see which diet is more suitable and effective for Malaysian FGID patients.

Participants will :

Be given either low FODMAP diet, Gentle FODMAP diet or Traditional Dietary Advice intervention and will be required to follow the intervention for two weeks.

Be required to provide stool and blood samples during baseline and intervention Record 4 day food diary and complete assessing questionnaires during baseline and intervention

DETAILED DESCRIPTION:
Functional Gastrointestinal Disorder (FGIDs), including irritable bowel syndrome (IBS) and functional dyspepsia (FD), are prevalent conditions that effects about 40% of world population and 21% of Malaysian population. They represent a significant health burden, impacting patients' quality of life. While the low FODMAP diet is effective in managing FGID around the western region, there is limited research done on comparing the impacts of diets with differing FODMAP content on symptom severity, quality of life, gut microbiota and gut barrier function of FGID patients in the Asian region as low FODMAP is restrictive. Therefore, conducting a randomised controlled trial is vital in measuring the effectiveness of diet with differing FODMAPs on FGID patients.

The objectives of this study are :

* To determine the effect of FODMAPs restriction on the gut microbiota abundance and diversity in FGID patients
* To determine the effect of FODMAPs restriction on gut barrier function after dietary intervention among FGID patients
* To determine the effect of FODMAPs restriction on the symptom severity, quality of life and psychological status in FGID patients

This study would be able to provide significant understanding of dietary management of FGID. Conducting this study would provide critical insights into the role of gut microbiota and gut barrier function in the pathophysiology of FGID, highlighting how dietary modulation can impact overall symptom management.

The study design involve screening and recruiting participants, followed by baseline data collection, randomisation, group allocation, and intervention with data collection.

First Visit (Day 1) During baseline, vital information such as socio demographic data will be gathered and FGID screening will be conducted using the ROME III Asian Diagnostic Questionnaire for Adults which consists of the Irritable Bowel Syndrome module and the Gastroduodenal Disorders module. A total of 5 questionnaires will be provide to the participants. These are Irritable Bowel Syndrome Severity Scale (IBS-SSS), Gastrointestinal Symptom Rating Scale (GSRS), Food avoidance and Dietary trigger questionnaire, Hospital Anxiety and Depression Scale (HADS), and the EQ-5D-5L questionnaire.

Body weight and composition of participants will be assessed using the Tanita Body Composition scale, whereas height of participants will be measured using a stadiometer. Dietary and FODMAPs will be estimated using a 4-day food diary (3 weekdays, 1 weekend). Additionally, blood sample will be collected from participants for further assessment. 10 ml blood will be drawn from each participant to detect serum biomarkers. Stool bottle will be provided to participants for stool collection upon the next visit. Stool collection is implemented to assess participants' gut integrity and gut microbiota. After concluding the baseline assessments, patients will be randomised into three groups. Groups A, B and C will follow a restricted FODMAP diet (LFD), Gentle FODMAP diet and traditional dietary advice (TDA), respectively. Participants will be randomly assigned to a study arm by a computer-generated randomisation program using the open-access website www.randomization.com at a ratio of 1:1:1.

Second Visit (Day 8) Participants will return their stool sample and completed diary. The diary will be assessed for completion, and the stool sample will be collected and frozen per protocol. Based on randomisation, participants in the LFD group will be provided with restricted FODMAP advice. In contrast, those in the GFD group will be given general healthy advice by dietitians/researchers trained in delivering the diet. Meanwhile, participants in the TDA group will be given an overall healthy dietary intervention and counselling. All three groups will be advised to follow their respective diets for two weeks. A food diary and another stool collection bottle will be provided.

Phone follow up (Day 15) A phone follow-up is scheduled after a week to remind participants to complete their food diary, answer any doubts or questions relating to their allocated intervention and subsequently plan their next visit.

Final visit (Day 22) Visit 3 will be scheduled after 2 weeks of intervention. Participants will return their stool samples, food diary, and questionnaire. They will also complete two symptom severity questionnaires, food avoidance and dietary trigger questionnaire, with questionnaires to assess quality of life and psychological status and provide a non-fasting blood sample. Additionally, participants in the LFD group will be provided advice on reintroduction. Those who have completed the study will be given an inconvenience allowance.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and above
* Able to provide informed consent
* Those with pre-existing irritable bowel syndrome (IBS) or functional dyspepsia (FD) or both screened by gastroenterologists
* Meet the ROME III- Asian criteria for FGID
* Able to communicate in Malay or English language

Exclusion Criteria:

* Pregnant or lactating women
* History declared by the participant of pre-existing gastrointestinal disorder, including but not limited to Inflammatory Bowel Disease, Coeliac Disease, Pancreatitis, Gallstone disease (biliary colic, cholecystitis), Diverticulitis
* Cancer of any kind
* Patients with reported history of previous resection of any part of the GI tract other than appendix or gall bladder, intestinal stoma
* Habitual use of opiate analgesics likely to alter bowel function e.g. morphine
* Use of antibiotics in the preceding two weeks and/or in the past one month
* Consumption of probiotics, prebiotics or fibre supplements in the past one month
* Enteral feeding or texture modified diet patients
* Those with cognitive impairment or severe mental disorder (Alzheimer's, schizophrenia, bipolar disorder. etc)
* Shift workers (e.g. Nurse, doctors)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-20 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Effect of FODMAP restrictions on Gut Microbiota Abundance and Diversity | Measurement before (Day 1) and after the diet (Day 22)
  16s RNA gene seqeuncing will be conducted on the stool samples at both baseline and post-intervention timelines. This test would target the microbial diversity by assessing the abdundance of key bacterial taxa.
Effect of FODMAP restrictions on Gut Barrier Function | Measurement before (Day 1) and after the diet (Day 22)
  The stool samples collected would be subjected to zonulin test and short-chain fatty acid quantification (SCFA) in order to assess gut barrier function of subjects at baseline and post-intervention timelines. Zonulin is a protein that reversibly modulates the intestinal permeability, while SCFA such as butyrate are by-products of the carbohydrate fermentation facilitated by gut microbiome that enhances the integrity of tight junction of the intestinal barrier

SECONDARY OUTCOMES:
Effect of 2 week FODMAP restrictions on Symptom Severity (IBS-SSS questionnaire) | Measurement before (Day 1) and after the diet (Day 22)
  Irritable Bowel Syndrome Symptom Severity Score (IBS-SSS) and Gastrointestinal Symptom Rating Scale (GSRS) will be filled out by subjects during baseline and post-intervention to assess symptom severity. For IBS-SSS, Four out of five items have visual analogue scales to describe the level of severity of abdominal pain, bloating or distension, disturbance of bowel habits and life impact of IBS symptoms. The level of severity will be categorised based on their total scores. A score of less than 25% is considered no pain, 25 to 50% is considered mild, 50 to 75% is considered moderate, and the score of 100% is very severe.
Effect of 2-week FODMAP restriction on Psychological Status | Measurement before (Day 1) and after the diet (Day 22)
  Hospital Anxiety and Depression Scale (HADS) will be filled out by subjects during baseline and post-intervention to assess symptom severity. This self-reported questionnaire contains 14 items that are scored on a 4-point Likert-type scale, ranging from 0 to 3, and are classified into two subscales measuring cognitive and emotional symptoms of depression (HADS-D) and anxiety (HADS-A). The total score on each subscale ranges from 0 to 21, and a higher score represents worse symptoms. A score equal to or greater than eight on either HADS-D or HADS-A is considered a 'possible case', and above 11 a 'probable case'.
Effect of 2-week FODMAP restriction on Quality of Life | Measurement before (Day 1) and after the diet (Day 22)
  European Quality of Life 5 Dimensions 5 Level Version Questionnaire (EQ-5D-5L) will be filled out by subjects during baseline and post-intervention to assess quality of life. This validated questionnaire consists of five items capturing different aspects of health, including mobility, self-care, ability to carry out usual activities, pain/discomfort and anxiety/depression. Each item has five levels of responses, where the minimum level being 'no problems' and maximum level being 'unable to do' things mentioned.
Effect of 2-week FODMAP restriction on Food Avoidance | Measurement before (Day 1) and after the diet (Day 22)
  A validated food avoidance and dietary trigger questionnaire will be filled out by subjects during baseline and post-intervention to assess food avoidance. This questionnaire is a 10-item tool in which question 1 is to identify dietary triggers of subjects. Question 2, 3, and 4 are follow up questions to assess bowel symptoms and dietary triggers. Question 5 that assess fear of eating, has a 6-point Likert scale, where the minimum point is 'Strongly Disagree' and the maximum point is 'Strongly Agree'.Question 6 assesses food avoidance behaviour using a 4-point Likert scale, where the minimum point is 'Never' and the maximum point is 'Always'. Questions 6,7,8,9 and 10 are used to assess patient's medical knowledge and medical history.
Effect of 2 week FODMAP restrictions on Anthropometry | Measurement before (Day 1) and after the diet (Day 22)
  The anthropometry parameters such as weight (in kilograms), height (in centimetres), and body mass index (BMI) (kg/m^2) will be assessed using standard protocols. To measure changes in body composition, weight, and BMI, the Body Impedance Analysis (BIA) will be used. Parameters such as percentage of body fat (%), visceral fat, muscle mass (kg) and total body water (%) will be measured.
FODMAP Intake Before and After Intervention | Measurement before (Day 1) and after the diet (Day 22)
  FODMAP intake will be estimated from the 4-day food diary (3 weekdays, 1 weekend) given to subjects both before intervention and after following 2-week intervention. FODMAP intake will be estimated using the Monash University Database
Effect of 2-week FODMAP restrictions on Symptom Severity (GSRS questionnaire) | Measurement before (Day 1) and after the diet (Day 22)
  The Gastrointestinal Symptom Rating Scale (GSRS) will be filled out by subjects during baseline and post-intervention to assess symptom severity. GSRS is 13 item questionnaire that are scored on a 7-point Likert scale, with the minimum point being 'no discomfort at all' and maximum value being 'very severe discomfort'.

CONTACTS AND LOCATIONS:
Overall Officials: Neoh Hui-Min, Assc. Prf, Study Chair — National University of Malaysia; Vanitha Mariappan, Dr, Study Chair — National University of Malaysia; Deborah Chia Hsin Chew, Dr, Study Chair — National University of Malaysia; Syaratul Dalina Yusoff, Dr, Study Chair — National University of Malaysia; Yee Xing You, Dr, Study Chair — National University of Malaysia; Yeong Yeh Lee, Prof, Study Chair — Universiti Sains Malaysia; Jaysrina Mahalinga Moorthy, Ms, Study Director — National University of Malaysia
Locations (1):
- Hospital Canselor Tuanku Muhriz Universiti Kebangsaan Malaysia, Jalan Yaacob Latif, Bandar Tun Razak, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No
We will not be sharing individual patient data to the trial registry to protect participant confidentiality, as institutional policies restrict such disclosure.

REFERENCES:
- [Background] Zia JK, Lenhart A, Yang PL, Heitkemper MM, Baker J, Keefer L, Saps M, Cuff C, Hungria G, Videlock EJ, Chang L. Risk Factors for Abdominal Pain-Related Disorders of Gut-Brain Interaction in Adults and Children: A Systematic Review. Gastroenterology. 2022 Oct;163(4):995-1023.e3. doi: 10.1053/j.gastro.2022.06.028. Epub 2022 Jun 16. PMID 35716771
- [Background] Murray K, Wilkinson-Smith V, Hoad C, Costigan C, Cox E, Lam C, Marciani L, Gowland P, Spiller RC. Differential effects of FODMAPs (fermentable oligo-, di-, mono-saccharides and polyols) on small and large intestinal contents in healthy subjects shown by MRI. Am J Gastroenterol. 2014 Jan;109(1):110-9. doi: 10.1038/ajg.2013.386. Epub 2013 Nov 19. PMID 24247211
- [Background] Melchior C, Desprez C, Riachi G, Leroi AM, Dechelotte P, Achamrah N, Ducrotte P, Tavolacci MP, Gourcerol G. Anxiety and Depression Profile Is Associated With Eating Disorders in Patients With Irritable Bowel Syndrome. Front Psychiatry. 2020 Jan 8;10:928. doi: 10.3389/fpsyt.2019.00928. eCollection 2019. PMID 31969841
- [Background] MacIntosh A, Heenan PE, Wright-McNaughton M, Frampton C, Skidmore P, Wall CL, Muir J, Talley NJ, Roy NC, Gearry RB. The relationship between fermentable carbohydrates and post-prandial bowel symptoms in patients with functional bowel disorders. Front Nutr. 2023 Feb 2;10:1060928. doi: 10.3389/fnut.2023.1060928. eCollection 2023. PMID 36819701
- [Background] Jang SH, Choi SC, Kim YS, Ryu HS, Lee SY, Bahk WM. Psychological Characteristics and Quality of Life of Patients with Upper and Lower Functional Gastrointestinal Disorders. J Clin Med. 2022 Dec 23;12(1):124. doi: 10.3390/jcm12010124. PMID 36614925
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Ghoshal UC, Gwee KA, Chen M, Gong XR, Pratap N, Hou X, Syam AF, Abdullah M, Bak YT, Choi MG, Gonlachanvit S, Chua AS, Chong KM, Siah KT, Lu CL, Xiong L, Whitehead WE. Development, Translation and Validation of Enhanced Asian Rome III Questionnaires for Diagnosis of Functional Bowel Diseases in Major Asian Languages: A Rome Foundation-Asian Neurogastroenterology and Motility Association Working Team Report. J Neurogastroenterol Motil. 2015 Jan 1;21(1):83-92. doi: 10.5056/jnm14045. PMID 25537673
- [Background] Chuah KH, Beh KH, Mahamad Rappek NA, Mahadeva S. The epidemiology and quality of life of functional gastrointestinal disorders according to Rome III vs Rome IV criteria: A cross-sectional study in primary care. J Dig Dis. 2021 Mar;22(3):159-166. doi: 10.1111/1751-2980.12975. PMID 33595169
- [Background] Burton Murray H, Riddle M, Rao F, McCann B, Staller K, Heitkemper M, Zia J. Eating disorder symptoms, including avoidant/restrictive food intake disorder, in patients with disorders of gut-brain interaction. Neurogastroenterol Motil. 2022 Aug;34(8):e14258. doi: 10.1111/nmo.14258. Epub 2021 Oct 24. PMID 34693609
- [Background] Black CJ, Drossman DA, Talley NJ, Ruddy J, Ford AC. Functional gastrointestinal disorders: advances in understanding and management. Lancet. 2020 Nov 21;396(10263):1664-1674. doi: 10.1016/S0140-6736(20)32115-2. Epub 2020 Oct 10. PMID 33049221
- [Background] Biesiekierski JR, Rosella O, Rose R, Liels K, Barrett JS, Shepherd SJ, Gibson PR, Muir JG. Quantification of fructans, galacto-oligosacharides and other short-chain carbohydrates in processed grains and cereals. J Hum Nutr Diet. 2011 Apr;24(2):154-76. doi: 10.1111/j.1365-277X.2010.01139.x. Epub 2011 Feb 21. PMID 21332832
- [Background] Bellini M, Tonarelli S, Nagy AG, Pancetti A, Costa F, Ricchiuti A, de Bortoli N, Mosca M, Marchi S, Rossi A. Low FODMAP Diet: Evidence, Doubts, and Hopes. Nutrients. 2020 Jan 4;12(1):148. doi: 10.3390/nu12010148. PMID 31947991
- [Background] Barrett JS, Gearry RB, Muir JG, Irving PM, Rose R, Rosella O, Haines ML, Shepherd SJ, Gibson PR. Dietary poorly absorbed, short-chain carbohydrates increase delivery of water and fermentable substrates to the proximal colon. Aliment Pharmacol Ther. 2010 Apr;31(8):874-82. doi: 10.1111/j.1365-2036.2010.04237.x. Epub 2010 Jan 22. PMID 20102355
- [Background] Atkins M, Zar-Kessler C, Madva EN, Staller K, Eddy KT, Thomas JJ, Kuo B, Burton Murray H. History of trying exclusion diets and association with avoidant/restrictive food intake disorder in neurogastroenterology patients: A retrospective chart review. Neurogastroenterol Motil. 2023 Mar;35(3):e14513. doi: 10.1111/nmo.14513. Epub 2023 Jan 4. PMID 36600490